CLINICAL TRIAL: NCT05450757
Title: A Prospective Multicentre Cohort Study of Acute ST-segment Elevation Myocardial Infarction
Brief Title: Shanghai ST-segment Elevation Myocardial Infarction Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, Director of Cardiology Department, Chief Physician, Ruijin Hospital
Other Study IDs: RJH-STEMI
Record Dates: First submitted 2022-07-02; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Acute Myocardial Infarction; Cardiac Remodelling; Heart Failure
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood samples at the time of pre-PCI, post-PCI, post-PCI 1 day, post-PCI 3days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ST-segment elevation myocardial infarction(STEMI) remains a major cause of morbidity and mortality worldwide, despite of the early reperfusion therapy, including fibrinolysis, primary percutaneous coronary intervention (PCI),and standardized medical treatment.To improve the prognosis of STEMI patients, the management in their hospitalization should be optimized, including improvements in risk stratification, more widespread use of an invasive strategy, implementation of care delivery systems prioritising immediate revascularisation through PCI (or fibrinolysis), advances in antiplatelet agents and anticoagulants, and greater use of secondary prevention strategies such as lipid-lowering therapy.

This study aims to standardized the management of STEMI patients and improve the prognosis of the STEMI patients.

DETAILED DESCRIPTION:
This study is a prospective cohort study. It aims to standardized the management of STEMI patients and improve the prognosis of the STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* ST elevation myocardial infarction
* Coronary angiography and percutaneous coronary intervention within 12 hours of symptom onset
* Capable and willing to provide informed conset and capable of completing study visits

Exclusion Criteria:

* Cardiovascular shock at admission
* Severe physical disability
* Active malignant tumors
* Active autoimmune diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is multi-center cohort study. Patients with acute ST elevation myocardial infarction undergo percutaneous coronary intervention within 12 hours of symptom onset at Ruijin Hospital, Minhang district Center Hospital, Yangpu district Center Hospital, Putuo district Center hospital,Jiading district Center Hospital, Fengxian district Center Hospital,and Shanghai Fifth people's Hospital, Shanghai, China are consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-09-12 (Actual); Primary Completion 2023-09-17 (Estimated); Study Completion 2024-09-17 (Estimated)

PRIMARY OUTCOMES:
MACE | 0-1 year
  Major adverse cardiovascular events(MACE) in one year follow-up
Left Ventricular Function | 1 month, 6month and 1 year
  Left ventricular end diastolic volume(LVEDV),Left ventricular end systolic volume(LVESE),Left ventricular ejection fraction(LVEF) changes within one year follow-up
Coronary angiography | 1 year
  The pathological changes in culprit vessels in 1 year

OTHER OUTCOMES:
Synchronized analysis of phonocardiogram and electrocardiogram | 1 day, 1 month, 6 months, 1 year
  Synchronized PCG and ECG data using a wearable cardiac monitoring patch

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wei Quan, M.D.,Ph.D., Study Chair — Ruijin Hospital; Tian Qi Zhu, M.D.,Ph.D., Study Chair — Ruijin Hospital; Xiao Xiang Yan, M.D.,Ph.D., Study Chair — Ruijin Hospital; Wen Li Zhang, M.D.,Ph.D., Study Chair — Ruijin Hospital; Run Du, M.D.,Ph.D., Study Chair — Ruijin Hospital; Ying Jia Xu, M.D.,Ph.D., Study Chair — Fudan University; Wei Hu, Study Chair — Shanghai Minhang District Central Hospital; Yimeng Zhou, Study Chair — Tongji University; Zongjun Liu, Study Chair — Shanghai Putuo District Central Hospital; Xiangdong Xu, Study Chair — Shanghai Jiading District Central Hospital; Zengyong Qiao, Study Chair — Shanghai Fengxian District Central Hospital
Locations (7):
- China (7):
  - Ruijin hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Fengxian District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Fifth People's Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Jiading District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Minhang District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Putuo District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Yangpu District Central Hospital, Shanghai, Shanghai Municipality